CLINICAL TRIAL: NCT07376447
Title: Confirmation of the Performance and Safety of the iNstroke 6F and 4F Thromboaspiration Catheter for the Treatment of Acute Ischemic Stroke
Brief Title: Evaluation of iNstroke Aspiration Catheters for Thrombectomy: a Multi-center Prospective Study
Acronym: iNDUO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: iVascular S.L.U. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iNDUO-01
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Ischemia; Thromboaspiration
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thromboaspiration using iNstroke 4F and/or iNstroke 6F aspiration catheter (Other): No comparator will be used in this clinical investigation as it is an exploratory study of a CE-marked medical device to be used within the scope of its intended purpose.
  Interventions: Device: Thromboaspiration catheter

INTERVENTIONS:
Device: Thromboaspiration catheter — Patients to undergo thromboaspiration with iNstroke 6F and/or 4F

SUMMARY:
Prospective, single-arm, multi-center study to confirm the performance and safety of the iNstroke 6F and 4F thromboaspiration catheter for the treatment of acute ischemic stroke

DETAILED DESCRIPTION:
This clinical investigation has been designed to generate further data demonstrating the safety and effectiveness of the iNstroke device as well as of the thrombectomy process for the treatment of large and medium vessel occlusions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age.
2. Able to be treated (i.e., defined by arterial puncture time) within 24 hours of symptom onset or last time seen well (LTSW).
3. Demonstrated occlusion in a large and/or medium vessel (carotid T, M1, proximal M2, M2-M3, A1, A2, A3, basilar artery, P1, P2, P3).
4. Baseline NIHSS score ≥6 assessed before the procedure.
5. Pre-morbid [xB13.1]stroke baseline mRS ≤ 2.
6. Subjects with an ASPECTS ≥ 6.
7. Informed consent signed by the subject or their representative, or notice of information, as per regulatory requirements, to collect the subject's data.
8. As applicable by French laws, the subject is affiliated to a health social security regimen or equivalent (only to be answered by French sites).

Exclusion Criteria:

1. Severe comorbidity and/or shortened life expectancy that will likely prevent improvement or follow up or that will render the procedure unlikely to benefit the patient.
2. Severe allergy to contrast media.
3. As applicable by French laws: breastfeeding women, persons deprived of their liberty by a judicial or administrative decision, or persons of full age who are the subject of a legal protection measure.
4. Patients with intracranial atherosclerotic occlusive disease or extra- or intracranial dissection.
5. Multiple Intracranial Occlusions
6. Known medical history of thrombocytopenia (Platelets <100,000).
7. Presence of intracerebral hemorrhage.
8. Significant mass effect and/or midline shift.
9. Evidence of intracranial tumor (except small meningioma).
10. Intracranial stenosis proximal to the occlusion.
11. Severe sustained hypertension (systolic pressure >185 mm Hg or diastolic pressure >110 mm Hg). Note: If blood pressure can be successfully reduced and maintained at an acceptable level by administering the medication recommended by the ESO (European Stroke Organisation) in its guidelines (also IV infusion of antihypertensives), the patient may be included.
12. Known or suspected cerebral vasculitis.
13. Known renal insufficiency with creatinine ≥3 mg/dl or Glomerular Filtration Rate (GFR) <30 mL/min.
14. Current participation in an interventional drug or device study that may confound the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-05-31 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recanalization Rate | Intra-procedure
  Recanalization rate with mTICI ≥2b in ≤3 revascularization passes using iNstroke Thrombus Extraction Aspiration Device aspiration catheter alone, or in conjunction with Stent Retriever.

CONTACTS AND LOCATIONS:
Locations (11):
- France (6):
  - CHU Bordeaux (H Pellegrin), Bordeaux
  - CHU Brest, Brest
  - CHU Lille, Lille
  - CHU Nancy, Nancy
  - APHP Pitié Salpétrière, Paris
  - CHU Strasbourg, Strasbourg
- Germany (5):
  - Klinikum Bremen Mitte, Bremen
  - Universität zu Köln, Cologne
  - Knappschaft Kliniken, Dortmund
  - UKE Hamburg, Hamburg
  - Klinikum Nürnberg, Nuremberg

IPD SHARING:
Plan to Share IPD: No